CLINICAL TRIAL: NCT01383200
Title: Comparison of 0.5% Tetracaine Drops Versus 2% Lidocaine Gel for Anesthetic Efficacy and Comfort in Patients Undergoing LASIK
Brief Title: Tetracaine Versus Lidocaine Gel for Anesthetic Effect and Comfort in Patients Undergoing LASIK
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: eyes that received gel had slightly thinner than intended flaps
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sonia Yoo, PROFESSOR, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20101016
Record Dates: First submitted 2011-06-13; First posted 2011-06-28 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: efficacy; comfort
MeSH Terms: conditions — Pain | interventions — Tetracaine; Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetracaine R/Lidocaine L (Active Comparator): Participant's Right or Left eye will receive 0.5% Tetracaine drop, at 10 minutes and 5 minutes, prior to LASIK.
  Interventions: Drug: Tetracaine drop; Drug: Lidocaine gel
- Tetracaine L/Lidocaine R (Active Comparator): Participant's Right or Left eye will receive 2% lidocaine gel, at 10 minutes and 5 minutes, prior to LASIK.
  Interventions: Drug: Tetracaine drop; Drug: Lidocaine gel

INTERVENTIONS:
Drug: Tetracaine drop — 0.5% Tetracaine Right eye / 2% Lidocaine Left eye
  Other Names: TetraVisc, Altacaine, AK-T-Caine and Pontocaine Ophthalmic
Drug: Lidocaine gel — 0.5% Tetracaine Left eye / 2% Lidocaine Right eye
  Other Names: Akten

SUMMARY:
In this study the investigators will be comparing two different types of anesthetic, a numbing eye drop and a numbing gel, to test if they are equally effective or if one has a better outcome in terms of the level of comfort you experience one hour and one day after your surgery. The two medications are commonly used and appear to be equally effective for other types of eye surgery, such as cataract surgery. This study will show if one type of anesthesia is preferred over another by patients getting LASIK. Before your LASIK procedure, you will be given a short questionnaire to determine the baseline comfort of your eyes. In the operating room, one type of anesthetic will be put in one eye, and the other medication will be put in the other eye. Which anesthetic you get in each eye will be chosen in a random way (similar to flipping a coin). After your LASIK surgery, the investigators will ask you if you felt more comfort in your right eye, your left eye, or if they were equal, and the investigators will ask you the same survey questions that were asked prior to your LASIK to get more details about your experience.

*Of note- the randomization being done is for which eye will be receiving the lidocaine and which eye will be receiving the tetracaine. Each patient will receive lidocaine in 1 eye and tetracaine in the other eye, the randomization is for each individual eye. This means, of 11 patients in our study, 22 eyes received treatment. 11 eyes received lidocaine and 11 eyes received tetracaine.

when we did our comparison, 11 values were used for lidocaine and 11 eyes were used for tetracaine, giving a total of 22 eyes. This is important to note since the randomization refers to EYE for each individual patient, and not for the patient (ie: participant means 1 eye, not 1 person in the descriptions below).

DETAILED DESCRIPTION:
Outcome measures involve comparing the right eye and left eye for severity of 12 different symptoms, that are recorded in severity on a 1-5 scale. A score of 1 means no symptoms and 5 means severe. The 12 measurements include sharp pain, dull ache, pain during movement, stinging sensation, itching, light sensitivity, watery eyes, dry eyes, sandy sensation, pressure sensation, decreased vision, and blurry vision.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers of age 18 years or greater

Exclusion Criteria:

* Previous reaction/allergy to the same drug class
* prior ocular surgery
* active facial injuries
* any active current ophthalmological disease
* history of diabetes
* any current non- Over The Counter pain medication
* inability to complete the questionnaire.
* Economically or educationally disadvantaged persons, Prisoners, or Children
* Patients with fluctuating or impaired decision-making capacity
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SONIA YOO, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

REFERENCES:
- [Derived] Shah NV, Vaddavalli PK, Chow JH, Roman JS, Shi W, Yoo SH. Prospective, double-masked, randomized trial comparing lidocaine gel to tetracaine drops in femtosecond laser-assisted LASIK. J Refract Surg. 2012 Oct;28(10):671-2. doi: 10.3928/1081597X-20121001-05. No abstract available. PMID 23061994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period is now over. Eligible patients included healthy patients undergoing bilateral LASIK surgery.
Groups:
- Tetracaine Right Eye / Lidocaine Left Eye: Each eye of the Subject was randomized using random number tables to receive either topical 0.5% tetracaine drops or 20% lidocaine gel
  11 eyes received 0.5% tetracaine drops.
- Tetracaine Left Eye / Lidocaine Right Eye: Each eye of the Subject was randomized using random number tables to receive either topical 0.5% tetracaine drops or 20% lidocaine gel
  11 eyes received 20% lidocaine gel.
Period: Overall Study
Arm/Group | Tetracaine Right Eye / Lidocaine Left Eye | Tetracaine Left Eye / Lidocaine Right Eye
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TetracaineRight Eye / LidocaineLeft Eye: 0.5% tetracaine drops Right eye /2% lidocaine gel Left eye
- TetracaineLeft Eye /LidocaineRight Eye: 0.5% tetracaine drops Left eye / 2% lidocaine gel Right eye
- Total: Total of all reporting groups
Arm/Group | TetracaineRight Eye / LidocaineLeft Eye | TetracaineLeft Eye /LidocaineRight Eye | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Participants Score on Pain Scale
Description: Do you have sharp pain in your eye? Pain will be assessed by units on a scale of 1-5: 1 means no symptoms, 2 means slight discomfort, 3 means mild discomfort, 4 means moderate discomfort, and 5 means severe discomfort
Time Frame: 1 hour (60minutes) post LASIK operation
Population: Five participants received tetracaine right eye and lidocaine left eye and six participants received lidocaine right eye and tetracaine left eye. A total of 22 eyes were analyzed for pain.
Measure: Mean (Standard Deviation); unit: Score on scale
Units Other Than Participants: eyes
Groups:
- Tetracaine: 0.5% tetracaine drops
- Lidocaine: 2% lidocaine gel
Arm/Group | Tetracaine | Lidocaine
Number analyzed (Participants) | 11 | 11
Number analyzed (eyes) | 11 | 11
Score on scale | 1.95 (.75) | 2.01 (.93)

ADVERSE EVENTS:
Groups:
- Tetracaine Right Eye / Lidocaine Left Eye: 0.5% Tetracaine drops Right eye / 2% Lidocaine Left eye
- Tetracaine Left Eye / Lidocaine Right Eye: 0.5% Tetracaine Left eye / 2% Lidocaine Right eye
Arm/Group | Tetracaine Right Eye / Lidocaine Left Eye | Tetracaine Left Eye / Lidocaine Right Eye
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No